CLINICAL TRIAL: NCT02349919
Title: Effect of Oral Procaterol on Chronic Persistent Cough Following Upper Respiratory Tract Infection: Double-Blind Randomized Placebo-Controlled Trial
Brief Title: Effect of Oral Procaterol on Postinfectious Persistent Cough
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Collaborators: Thai Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 002-TOI-2014-01
Record Dates: First submitted 2015-01-26; First posted 2015-01-29 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Cough
Keywords: postinfectious cough, postviral cough
MeSH Terms: conditions — Cough | interventions — Procaterol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Procaterol (Experimental): Procaterol 25 micrograms/tablet, 1 tablet twice daily for 4 weeks
  Interventions: Drug: Procaterol
- Placebo (Placebo Comparator): Placebo twice daily for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Procaterol — Procaterol 25 micrograms/tablet, 1 tablet twice daily for 4 weeks
  Other Names: procaterol hydrochloride
  Arms: Procaterol
Drug: Placebo — Placebo twice daily for 4 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effectiveness of oral procaterol in treatment of non-asthmatic patients who suffer from persistent cough following upper respiratory tract infection (URTI).

DETAILED DESCRIPTION:
Persistent cough following upper respiratory tract infection (URTI) is a common problem in the clinical practice, namely post-infectious cough. The potential mechanisms are viral-induced airway epithelial damage that leads to 1) airway hyperresponsiveness and airway narrowing, 2) increase in vascular permeability resulting in airway edema, and 3) activation of inflammatory mediators from inflammatory cells resulting in airway smooth muscle contraction. It is usually spontaneously resolved, although various therapeutic trials have been used with unpredictable results. Regarding to bronchodilators, inhaled ipratropium was effective in reducing cough symptom in a small study (N=14). We conduct a double-blind randomized placebo-controlled trial to investigate the effectiveness of oral procaterol, as a bronchodilator, in non-asthmatic adult patients suffering from persistent cough post URTI.

Eligible patients who have cough lasting longer than 3 weeks post URTI with normal spirometry will be randomized to receive either placebo or procaterol (25 microgram twice daily) for 4 weeks.

The primary outcome is cough symptom score using Leicester cough questionnaire (LCQ). The secondary outcomes are pulmonary function tests (spirometry, impulse oscillometry) and exhaled nitric oxide and quality of life (SF-36). All outcomes are measured at baseline, 2 weeks, and 4 weeks. Bronchoprovocation test with methacholine is performed at baseline and 4 weeks to determine the provocative concentration of methacholine that induces falling of FEV1 >or =20%. Adverse events will be recorded every visit.

Data analysis will be in both intention-to-treat and per-protocol fashion. A linear mixed-effect regression model will be applied to assess treatment effect on LCQ score, SF-36, and lung function. Within-subject variation will be fitted in the model as random effects whereas the treatment will be considered as a fixed effect. Time at measurement (i.e., 2- and 4-week) will also be included in the mixed model by treating it as fixed-effect. Marginal treatment effects between treatments and time will be then estimated and compared.

ELIGIBILITY:
Inclusion Criteria:

1. Having persistent cough that lasts longer than 3 weeks following URTI
2. Currently being a non-smoker
3. Having normal spirometry (FEV1>or= 80% predicted)
4. Obtain consent form

Exclusion Criteria:

1. Having cough more than 8 weeks
2. Having history of allergic or intolerance to β2 agonist
3. Having diagnosis of asthma by physicians
4. Presence of wheeze or rhonchi on physical examination
5. Having radiographic evidence of pneumonia, tuberculosis or sinusitis
6. Having significant gastroesophageal reflux symptoms suggested by GERD-Q questionnaire (GERD-Q score > 8)
7. Currently taking ACE-inhibitor
8. Being active smokers
9. Refuse to participate in the study

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Total score from Leicester cough questionnaire | up to 4 weeks

SECONDARY OUTCOMES:
Quality of life score from SF-36 | 2 weeks and 4 weeks
Spirometric parameters (FEV1, Forced expiratory flow between 25% and 75% of vital capacity; FEF25-75%) | 2 weeks and 4 weeks
Impulse oscillometry parameters (airway resistance at 5 Hz, and 20 Hz, difference of airway resistance at 5 Hz and 20 Hz) | 2 weeks and 4 weeks
Provocative concentration of methacholine that induces falling of FEV1 > or= 20% (PC20) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prapaporn Pornsuriyasak, M.D., Principal Investigator — Pulmonary and Critical Care, Department of Medicine, Ramathibodi Hospital, Mahidol University; Theerasuk Kawamatawong, M.D., Study Chair — Pulmonary and Critical Care, Department of Medicine, Ramathibodi Hospital, Mahidol University; Poungrat Thungtitigul, M.D., Study Director — Pulmonary and Critical Care, Department of Medicine, Ramathibodi Hospital, Mahidol University
Locations (1):
- Ramathibodi Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Hegele RG, Hayashi S, Hogg JC, Pare PD. Mechanisms of airway narrowing and hyperresponsiveness in viral respiratory tract infections. Am J Respir Crit Care Med. 1995 May;151(5):1659-64; discussion 1664-5. doi: 10.1164/ajrccm.151.5.7735630.
- [Background] Blair HT, Greenberg SB, Stevens PM, Bilunos PA, Couch RB. Effects of rhinovirus infection of pulmonary function of healthy human volunteers. Am Rev Respir Dis. 1976 Jul;114(1):95-102. doi: 10.1164/arrd.1976.114.1.95. PMID 180856
- [Background] Empey DW, Laitinen LA, Jacobs L, Gold WM, Nadel JA. Mechanisms of bronchial hyperreactivity in normal subjects after upper respiratory tract infection. Am Rev Respir Dis. 1976 Feb;113(2):131-9. doi: 10.1164/arrd.1976.113.2.131. PMID 1247226
- [Background] Nadel JA. Some epithelial metabolic factors affecting airway smooth muscle. Am Rev Respir Dis. 1988 Dec;138(6 Pt 2):S22-3. doi: 10.1164/ajrccm/138.6_Pt_2.S22. PMID 3059901
- [Background] Barnett K, Jacoby DB, Nadel JA, Lazarus SC. The effects of epithelial cell supernatant on contractions of isolated canine tracheal smooth muscle. Am Rev Respir Dis. 1988 Oct;138(4):780-3. doi: 10.1164/ajrccm/138.4.780. PMID 3202451
- [Background] Ida S, Hooks JJ, Siraganian RP, Notkins AL. Enhancement of IgE-mediated histamine release from human basophils by viruses: role of interferon. J Exp Med. 1977 Apr 1;145(4):892-906. doi: 10.1084/jem.145.4.892. PMID 67173
- [Background] Busse WW, Swenson CA, Borden EC, Treuhaft MW, Dick EC. Effect of influenza A virus on leukocyte histamine release. J Allergy Clin Immunol. 1983 Apr;71(4):382-8. doi: 10.1016/0091-6749(83)90066-0. PMID 6187791
- [Background] Chonmaitree T, Lett-Brown MA, Grant JA. Respiratory viruses induce production of histamine-releasing factor by mononuclear leukocytes: a possible role in the mechanism of virus-induced asthma. J Infect Dis. 1991 Sep;164(3):592-4. doi: 10.1093/infdis/164.3.592. PMID 1714484
- [Background] Volovitz B, Faden H, Ogra PL. Release of leukotriene C4 in respiratory tract during acute viral infection. J Pediatr. 1988 Feb;112(2):218-22. doi: 10.1016/s0022-3476(88)80058-1. PMID 3339502
- [Background] SALEM H, AVIADO DM. ANTITUSSIVE DRUGS, WITH SPECIAL REFERENCE TO A NEW THEORY FOR THE INITATION OF THE COUGH REFLEX AND THE INFLUENCE OR BRONCHODILATORS. Am J Med Sci. 1964 May;247:585-600. No abstract available. PMID 14158494
- [Background] Hueston WJ. A comparison of albuterol and erythromycin for the treatment of acute bronchitis. J Fam Pract. 1991 Nov;33(5):476-80. PMID 1940815
- [Background] Pornsuriyasak P, Charoenpan P, Vongvivat K, Thakkinstian A. Inhaled corticosteroid for persistent cough following upper respiratory tract infection. Respirology. 2005 Sep;10(4):520-4. doi: 10.1111/j.1440-1843.2005.00732.x. PMID 16135178
- [Background] Fuller RW, Jackson DM. Physiology and treatment of cough. Thorax. 1990 Jun;45(6):425-30. doi: 10.1136/thx.45.6.425. No abstract available. PMID 2203180
- [Background] Holmes PW, Barter CE, Pierce RJ. Chronic persistent cough: use of ipratropium bromide in undiagnosed cases following upper respiratory tract infection. Respir Med. 1992 Sep;86(5):425-9. doi: 10.1016/s0954-6111(06)80010-7. PMID 1462022
- [Background] Fujimura M, Sakamoto S, Kamio Y, Bando T, Kurashima K, Matsuda T. Effect of inhaled procaterol on cough receptor sensitivity to capsaicin in patients with asthma or chronic bronchitis and in normal subjects. Thorax. 1993 Jun;48(6):615-8. doi: 10.1136/thx.48.6.615. PMID 8346491
- [Background] Eldon MA, Battle MM, Coon MJ, Nordblom GD, Sedman AJ, Colburn WA. Clinical pharmacokinetics and relative bioavailability of oral procaterol. Pharm Res. 1993 Apr;10(4):603-5. doi: 10.1023/a:1018966506819. PMID 8483846
- [Background] Raj AA, Pavord DI, Birring SS. Clinical cough IV:what is the minimal important difference for the Leicester Cough Questionnaire? Handb Exp Pharmacol. 2009;(187):311-20. doi: 10.1007/978-3-540-79842-2_16. PMID 18825348
- [Background] Becker LA, Hom J, Villasis-Keever M, van der Wouden JC. Beta2-agonists for acute bronchitis. Cochrane Database Syst Rev. 2011 Jul 6;(7):CD001726. doi: 10.1002/14651858.CD001726.pub4. PMID 21735384